CLINICAL TRIAL: NCT06571617
Title: Retrograde Intrarenal Surgery Versus Mini-Percutaneous Nephrolithotomy for Treatment of Medium Size Pediatric Renal Stones (10-20millimeters). A Randomized Controlled Trial
Brief Title: F-URS and Mini PCNL for Pediatric Urolithiasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ramy Elbaz, assistant lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22.08.684
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Intervention Model Description: Patients will be randomized using computer-generated random tables in a 1:1 ratio to be allocated to one of two groups, the first group will undergo mini-PNL, and the second group will undergo RIRS.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini PCNL (mini percutaneous nephrolithotomy) (Active Comparator): Under general anesthesia, a 5/ 6 Fr ureteric catheter will be placed in the pelvicalyceal system. then the patient is turned to the prone position. A puncture will be done using an 18 G needle under fluoroscopy guidance. The tract will be dilated up to 15 F and then a sheath will be placed. A 12 F nephoscope (MIP-M, Karl Storz Endoscopy, Tuttlingen, Germany) will be used. Stone fragmentation will be performed using holmium YAG Laser energy. Then, Fragments will be evacuated using vacuum cleaner effect, tipless basket, or 5 FR stone forceps for stone analysis. A nephrostomy tube 12 Fr will be fixed at the end of the procedure.
  Interventions: Procedure: Mini PCNL (mini percutaneous nephrolithotomy)
- RIRS (retrograde intrarenal surgery/ flexible URS) (Active Comparator): Under general anesthesia, the children will be placed in the lithotomy position . Cystoscopy or rigid ureteroscopy will be performed to place a hydrophilic guidewire to the renal pelvis under fluoroscopic guidance. After passing a 0.035/0.038-inch safety guidewire into the renal pelvis, a ureteral access sheath will be placed (9.5/11.5 Fr, 35 cm) will be used according to the surgeon preference. . RIRS will be performed using a single use digital Flexible ureteroscopy . A manual irrigation pump system will be used to hydro dilate the ureter during ureteroscopy. The stones will be fragmented with a holmium:YAG laser until they will be deemed small enough to pass spontaneously. Some residual fragments will be removed by tipless nitinol basket for stone analysis. A double-J stent OR URETERIC CATHETER will be placed at the end of the procedure based on surgeon's decision. .
  Interventions: Procedure: RIRS (retrograde intrarenal surgery/ flexible URS)

INTERVENTIONS:
Procedure: Mini PCNL (mini percutaneous nephrolithotomy) — half of the cases will be treated using mini PCNL
  Arms: Mini PCNL (mini percutaneous nephrolithotomy)
Procedure: RIRS (retrograde intrarenal surgery/ flexible URS) — THE OTHER HALF WILL BE TRAETED USING Flexible URS
  Arms: RIRS (retrograde intrarenal surgery/ flexible URS)

SUMMARY:
To compare RIRS versus mini-perc PNL in the management of medium size pediatric renal stones (10-20 mm) through a RCT.

DETAILED DESCRIPTION:
Pediatric urolithiasis has become a major health problem, especially in the developing countries. It is a well-known risk factor for renal impairment and end-stage kidney disease (ESKD). Also, it's associated with a bad quality of life (Qol) for both parents and child. Children represent 2-3% of the total population of stone-formers. Similar to adult urolithiasis, the prevalence of pediatric stones is widely variable in different parts of the world. it changes with sex, race, geographical and climatic factors.

Renal stones in pediatric patients are usually caused by an underlying disorder, such as anatomical and metabolic anomalies or recurrent urinary tract infections, So, children with renal stones are at higher risk for recurrence and multiple interventions on the kidney Over the last decades, the management of pediatric urolithiasis had been replaced by less invasive endourological procedures and the role of open surgeries had been greatly subsided. According to the last guidelines from the European Association of Urology (EAU) and the American urological association (AUA), the standard treatment of renal stones between1-2 cm is shockwave lithotripsy (SWL), percutaneous nephrolithotomy (PNL) and retrograde intrarenal surgery (RIRS). However, the first choice between these modalities is still controversial until now.

SWL is one of the most effective treatment options for pediatric stones, however, its long-term effect on developing kidneys is not clear yet. Also, its efficacy decreases significantly with increasing stone size and multiplicity. The requirement for multiple sessions and the need for general anesthesia in children are other drawbacks of this procedure.

PNL has significantly higher stone-free rates (SFR) and lower requirements for auxiliary procedures compared with SWL. This trend is further promoted by the introduction of miniaturized PNL (mini-perc), which is postulated to be less invasive compared with standard PNL because of the miniaturized instruments. However, PNL may present problems in children, despite modifications, such as the "mini-perc," because of the small size and mobility of the pediatric kidney, friable renal parenchyma, and the small size of the collecting system.

On the other hand, the quality of flexible ureteroscopy and endoscopic instruments showed an outstanding development over the last years which made RIRS a feasible option for pediatric renal stones. Experience suggests that flexible ureteroscopy has a lower risk of kidney damage and bleeding. However, the disadvantage of RIRS in children includes the need toindwell double-J stent in advance, the risk of ureteral injury, and the high cost of equipment purchase and maintenance, which may limit the application of RIRS in children with upper urinary tract calculi.

Until now, there is a few number of randomized trials compared mini-perc PNL versus RIRS for pediatric renal stones. SO, there is no clear evidence for the superiority of one option over the other regarding stone- free rate, complication rate, auxiliary procedures, and second sessions.

Recently, a new Trifecta tool which includes stone-free status in a single session without complications was set in motion to help standard reporting of the outcome of stone intervention in line with assessing its efficacy and safety.

In the present study, we will try to overcome the limitations of the previous studies by designing a prospective randomized controlled trial (RCT). To the best of our knowledge, the present study is the first RCT comparing mini-perc PNL versus RIRS for the management medium -size renal stones (10-20mm) in children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12 years or younger
* American society of anesthesia (ASA) score I or II.
* Renal stone measured between 10-20 mm.
* An informed consent obtained from their parents

Exclusion Criteria:

* Bleeding tendency
* Active urinary tract infection (UTI).
* Renal anatomical abnormalities (ectopic kidney, horseshoe kidney, ADPCK).
* Skeletal deformities
* Concomitant ureteric stone or stricture.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-04-05 (Estimated)

PRIMARY OUTCOMES:
the primary outcome, the stone-free rate | at 4 weeks postoperatively
  no evidence of any residual fragment by NCCT or KUB or clinical insignificant residual fragments (CIRF) ≤ 4 mm in maximum diameter in a single session within the first month postoperatively.

SECONDARY OUTCOMES:
The Secondary outcomes, perioperative parameters | intraoperative and first day postoperatively
  intraoperative complications, operation time in minutes, fluoroscopy time in seconds, lasing time in seconds, laser energy in joles, hemoglobin deficit, postoperative complications, hospital stay in days

OTHER OUTCOMES:
the tertiary outcome. post operative pain score | at first day post operative
  assessment of pain at postoperative day 1 (PODI), For children < 7.5 years, we will use the validated Arabic version of Wong-Baker FACES scale (WBF). For older children, we will use the validated Arabic version of visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Ramy F Elbaz, Principal Investigator — Mansoura University
Locations (1):
- Urology and nephrology center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
plan to share the surgical techniques in both arms, post operative outcomes and statistics results
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after 4 months for 6 months
Access Criteria: via email: ramifrag7@gmail.com